CLINICAL TRIAL: NCT03631303
Title: Post-Extrasystolic Potentiation as a Predictor of Ventricular Arrhythmias
Acronym: A PRIORY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Cornelis P. Allaart, Principal Investigator, Amsterdam UMC, location VUmc
Other Study IDs: 2018.246
Record Dates: First submitted 2018-08-12; First posted 2018-08-15 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Post-extrasystolic Potentiation (PESP); Ventricular Tachycardia
Keywords: Implantable cardioverter defibrillator; Post-extrasystolic Potentiation; Sudden Cardiac Death
MeSH Terms: conditions — Tachycardia, Ventricular; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- ICD patients with ATP/shock: 10 primary prevention 2-chamber ICD patients (LVEF <35 percent) who received appropriate ICD therapy during follow-up.
  Interventions: Device: Cardiac stimulation through the device leads
- ICD patients without ATP/Shock: 10 primary prevention 2-chamber ICD patients (LVEF <35 percent) who were free from appropriate ICD therapy during follow-up.
  Interventions: Device: Cardiac stimulation through the device leads
- Pacemaker-patients: 10 2-chamber pacemaker-patients (LVEF >50%).
  Interventions: Device: Cardiac stimulation through the device leads

INTERVENTIONS:
Device: Cardiac stimulation through the device leads — During scheduled device replacement extra-systolic beats with various extrasystolic and post-extrasystolic coupling intervals will be evoked by electrical stimulation via the right atrial and ventricular device leads of the patient. Throughout the stimulation study blood pressure will be measured non-invasively using a finger arterial blood pressure photoplethysmographic device and a continuous electrocardiogram will be recorded.

SUMMARY:
Background: Patients at increased risk for sudden cardiac death (SCD) may receive an implantable cardioverter defibrillator (ICD). The primary criterion for a primary prevention ICD implantation is a left ventricular ejection fraction (LVEF) below 35%, but refinement of ICD criteria is important since only a small proportion of ICD patients receives appropriate device therapy (ATP or a shock) during follow-up. Post-extrasystolic potentiation (PESP) may be a new risk marker for SCD. PESP is defined as a temporary increase in contractility that follows an extrasystolic beat (ESB) and is associated with myocardial calcium handling. In heart failure, changes in calcium homeostasis may lead to afterdepolarisations and thus predispose for SCD. PESP can be measured indirectly and non-invasively as post-extrasystolic blood pressure potentiation (PESP-BP). Abnormal PESP-BP was previously found to be an independent predictor of increased mortality in post-myocardial infarction patients with a reduced LVEF. However, it is unknown if this increased mortality in heart failure patients with abnormal PESP-BP is caused by an increased risk of SCD.

Hypothesis: The investigators hypothesize that PESP-BP might be a new predictor of the occurrence of SCD, and can be used to enhance patient selection for primary prevention ICD therapy.

Design: During scheduled device replacement ESB with various extrasystolic and post-extrasystolic coupling intervals will be evoked by electrical stimulation via the right atrial and ventricular device leads of the patient. Throughout the stimulation study blood pressure will be measured non-invasively a continuous electrocardiogram will be recorded. Either before or after the procedure, patients will undergo a 30-minutes assessment of spontaneous ESB, again with blood pressure and ECG recordings.

Study population: 30 patients who are scheduled for device replacement or reposition, are eligible for this study; (1) 10 ICD patients who previously received appropriate device therapy (ADT); (2) 10 ICD patients who are free from ADT and (3) 10 dual-chamber pacemaker patients (control group).

Outcomes: (1) Evoked PESP-BP (i.e. blood pressure differences between baseline, ESB and post-ESB); (2) Spontaneous PESP-BP (i.e. blood pressure differences between baseline, ESB and post-ESB); (3) Timing parameters (in ms): the basic cycle length interval; Extra-systolic interval (ESI); Post-extrasystolic interval (PESI).

ELIGIBILITY:
Inclusion Criteria:

* Implanted with a dual-chamber device
* For ICD patients: a LVEF ≤35%, measured recently
* For Pacemaker patients: a LVEF > 50% measured both recently
* A device follow-up of at least one year must be available
* Optimal (stable) medical therapy
* Sinus rhythm

Exclusion Criteria:

* Age <18 or incapacitated adult
* Unknown left ventricular function prior to device implantation
* Patients unwilling to participate
* Documented atrial fibrillation
* Second or third degree atrioventricular (AV) conduction disorders;
* Patients with a cardiac resynchronization therapy (CRT-D) or one-chamber device
* Hypertrophic cardiomyopathy
* Conditions with insufficient blood flow to the fingers, e.g. M. Raynaud or conditions with extreme vasoconstriction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients who are scheduled for device replacement or reposition, are eligible for this study; (1) 10 ICD patients who previously received appropriate device therapy (ATP/shock); (2) 10 ICD patients who are free from ADT and (3) 10 dual-chamber pacemaker patients (control group)
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Evoked PESP-BP | Measured during stimulation protocol
  blood pressure differences between baseline, extrasystolic beat (ESB) and post-ESB
Spontaneous PESP-BP | Measured in rest, without cardiac stimulation with spontaneous ESB
  blood pressure differences between baseline, extrasystolic beat (ESB) and post-ESB

CONTACTS AND LOCATIONS:
Overall Officials: Cornelis P. Allaart, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU university medical center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Steger A, Sinnecker D, Barthel P, Muller A, Gebhardt J, Schmidt G. Post-extrasystolic Blood Pressure Potentiation as a Risk Predictor in Cardiac Patients. Arrhythm Electrophysiol Rev. 2016 May;5(1):27-30. doi: 10.15420/aer.2016.14.2. PMID 27403290
- [Background] Sinnecker D, Dirschinger RJ, Barthel P, Muller A, Morley-Davies A, Hapfelmeier A, Dommasch M, Huster KM, Hasenfuss G, Laugwitz KL, Malik M, Schmidt G. Postextrasystolic blood pressure potentiation predicts poor outcome of cardiac patients. J Am Heart Assoc. 2014 Jun 3;3(3):e000857. doi: 10.1161/JAHA.114.000857. PMID 24895163